CLINICAL TRIAL: NCT02192827
Title: Single Dose Dexamethasone is as Effective as Two Doses in Mild to Moderate Pediatric Asthma Exacerbations in the Emergency Department
Brief Title: Use of Dexamethasone in Pediatric Asthma Exacerbations
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University at Buffalo (Other)
Responsible Party: Principal Investigator, Meghan Martin, Pediatric Emergency Medicine Attending Physician, University at Buffalo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 647430-4
Record Dates: First submitted 2014-07-11; First posted 2014-07-17 (Estimated); Results first posted 2023-03-30 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Asthma
Keywords: Pediatric; Asthma; Exacerbation; Dexamethasone
MeSH Terms: conditions — Asthma | interventions — dexamethasone 21-phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Single Dose Dexamethasone (Experimental): 0.6 mg/kg of Dexamethasone Sodium Phosphate Injection 10mg/1ml given with equivalent volume of cherry syrup given orally once
  Interventions: Drug: Dexamethasone Sodium Phosphate Injection
- Two Dose Dexamethasone (Experimental): 0.6 mg/kg of Dexamethasone Sodium Phosphate Injection 10mg/1ml given with equivalent volume of cherry syrup given orally once in the Emergency Department (ED), followed by another dose of dexamethasone at home, which will be prescribed from the ED. The second dose will be the same dosage, but will be prescribed and may be pill or liquid form.
  Interventions: Drug: Dexamethasone Sodium Phosphate Injection

INTERVENTIONS:
Drug: Dexamethasone Sodium Phosphate Injection

SUMMARY:
The purpose of this study is to compare the efficacy of a single dose of dexamethasone vs. two doses of dexamethasone in mild and moderate asthma exacerbations pediatric patients.

DETAILED DESCRIPTION:
The emergency department (ED) physician will follow the standard asthma care path to manage a pediatric asthma patient whether the patient meets study criteria or not. Patients' legal guardian will be approached for consent if patient meets the study criteria. Once the consent is obtained, the patient will be randomized into one of the two study groups according to a randomization table generated by a statistician. The first group will receive a single dose of dexamethasone sodium phosphate injection (0.6 mg/kg with max of 16 mg) mixed with equivalent volume of cherry syrup given orally in the ED. The second group will receive a first dose of dexamethasone with cherry syrup (also 0.6 mg/kg with max of 16 mg) in the ED, and a second dose will be prescribed to the patient at home on the day following the ED visit. This dose will be the same dosage of dexamethasone, but may be a pill or liquid form. Patients will continue their previously prescribed asthma regimen and albuterol as needed. Children who vomit the steroids in the ED will be re-dosed. Children who vomit the steroid a second time will be excluded from the study.

2. Data collection. Demographic information such as age, race, duration of asthma symptoms, number of previous hospitalizations, and current medication will be collected on an ED data collection form. Pertinent exam findings such as patient's vital signs, pulse oximetry, Pediatric asthma severity score (PAS), patient asthma severity self-assessment sheets (PSAS), and ED treatment will also be collected on an ED data collection form.

After discharge from the ED, patients will be instructed to complete the PSAS on a daily basis for 5 days. The data will be documented on a home patient self-assessment sheet by the legal guardian. The investigators will train the legal guardians on how to complete the PSAS in the ED.

3. Phone follow-up All patients will be contacted by phone by a research assistant 5 days after the ED visit. Information collected during the phone interview will include PSAS, unexpected visits to medical providers (ED, primary care or urgent care) for asthma symptoms, school days missed due to asthma exacerbation, length of time symptoms persisted, compliance with the recommended steroid regimen, vomiting, other side effects or medication administration problems caused by the steroids.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 2 to 20 years, from all race and ethnicity groups, with a known history of asthma who present to the Emergency Department of Women and Children's Hospital of Buffalo with an acute exacerbation of mild or moderate asthma are potentially eligible for the study. Patients with severe asthma exacerbations will require intravenous steroid therapy, therefore, they will not be enrolled in the study. The investigators plan to enroll patients from winter of 2014 to fall 2016.

History of asthma is defined by physician diagnosis of at least 1 prior episode of wheezing which responded to beta agonist medication.

Mild asthma is defined as: Pediatric Asthma Score (PAS) of 5 to 7; Moderate asthma is defined as: PAS of 8 to 11; Severe asthma is defined as: PAS of 12 or more.

Exclusion Criteria:

* Children who have one of the following conditions will be excluded from the study: are less than 2 years of age, have signs of severe exacerbation (Pediatric Asthma Score of more than 11), have used oral steroids in the last 2 weeks, have chronic lung disease (e.g., cystic fibrosis), have been given IV solumedrol, or vomit two doses of dexamethasone in emergency department.

Ages: 2 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 318 (Actual)
Dates: Start 2015-04; Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Meghan E Martin, MD, Principal Investigator — Johns Hopkins All Children's Hospital
Locations (1):
- Women and Children's Hospital Of Buffalo, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Akinbami LJ, Simon AE, Rossen LM. Changing Trends in Asthma Prevalence Among Children. Pediatrics. 2016 Jan;137(1):1-7. doi: 10.1542/peds.2015-2354. Epub 2015 Dec 28. PMID 26712860
- [Background] National Asthma Education and Prevention Program. Expert Panel Report 3 (EPR-3): Guidelines for the Diagnosis and Management of Asthma-Summary Report 2007. J Allergy Clin Immunol. 2007 Nov;120(5 Suppl):S94-138. doi: 10.1016/j.jaci.2007.09.043. PMID 17983880
- [Background] Chapman KR, Verbeek PR, White JG, Rebuck AS. Effect of a short course of prednisone in the prevention of early relapse after the emergency room treatment of acute asthma. N Engl J Med. 1991 Mar 21;324(12):788-94. doi: 10.1056/NEJM199103213241202. PMID 1997850
- [Background] Rachelefsky G. Treating exacerbations of asthma in children: the role of systemic corticosteroids. Pediatrics. 2003 Aug;112(2):382-97. doi: 10.1542/peds.112.2.382. PMID 12897291
- [Background] Scarfone RJ, Fuchs SM, Nager AL, Shane SA. Controlled trial of oral prednisone in the emergency department treatment of children with acute asthma. Pediatrics. 1993 Oct;92(4):513-8. PMID 8414819
- [Background] Zoorob RJ, Cender D. A different look at corticosteroids. Am Fam Physician. 1998 Aug;58(2):443-50. PMID 9713398
- [Background] Cronin J, Kennedy U, McCoy S, An Fhaili SN, Crispino-O'Connell G, Hayden J, Wakai A, Walsh S, O'Sullivan R. Single dose oral dexamethasone versus multi-dose prednisolone in the treatment of acute exacerbations of asthma in children who attend the emergency department: study protocol for a randomized controlled trial. Trials. 2012 Aug 21;13:141. doi: 10.1186/1745-6215-13-141. PMID 22909281
- [Background] Karaman M, Ilhan AE, Dereci G, Tek A. Determination of optimum dosage of intraoperative single dose dexamethasone in pediatric tonsillectomy and adenotonsillectomy. Int J Pediatr Otorhinolaryngol. 2009 Nov;73(11):1513-5. doi: 10.1016/j.ijporl.2009.06.001. Epub 2009 Jul 10. PMID 19801100
- [Background] Qureshi F, Zaritsky A, Poirier MP. Comparative efficacy of oral dexamethasone versus oral prednisone in acute pediatric asthma. J Pediatr. 2001 Jul;139(1):20-6. doi: 10.1067/mpd.2001.115021. PMID 11445789
- [Background] Greenberg RA, Kerby G, Roosevelt GE. A comparison of oral dexamethasone with oral prednisone in pediatric asthma exacerbations treated in the emergency department. Clin Pediatr (Phila). 2008 Oct;47(8):817-23. doi: 10.1177/0009922808316988. Epub 2008 May 8. PMID 18467673
- [Background] Keeney GE, Gray MP, Morrison AK, Levas MN, Kessler EA, Hill GD, Gorelick MH, Jackson JL. Dexamethasone for acute asthma exacerbations in children: a meta-analysis. Pediatrics. 2014 Mar;133(3):493-9. doi: 10.1542/peds.2013-2273. Epub 2014 Feb 10. PMID 24515516
- [Background] Kelly CS, Andersen CL, Pestian JP, Wenger AD, Finch AB, Strope GL, Luckstead EF. Improved outcomes for hospitalized asthmatic children using a clinical pathway. Ann Allergy Asthma Immunol. 2000 May;84(5):509-16. doi: 10.1016/S1081-1206(10)62514-8. PMID 10831004
- [Background] Chang AB, Clark R, Sloots TP, Stone DG, Petsky HL, Thearle D, Champion AA, Wheeler C, Acworth JP. A 5- versus 3-day course of oral corticosteroids for children with asthma exacerbations who are not hospitalised: a randomised controlled trial. Med J Aust. 2008 Sep 15;189(6):306-10. doi: 10.5694/j.1326-5377.2008.tb02046.x. PMID 18803532

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients presenting with asthma symptoms to a single pediatric emergency department
Pre-assignment Details: Excluded 10 Patients:
  Previously enrolled into the study: 2 Admitted to the PICU (pediatric intensive care unit): 5 Required IV steroids in the Emergency Dept: 1 Steroid use within the last 2 weeks: 1 Excessive vomiting in the Emergency Dept: 1
Groups:
- Single Dose Dexamethasone: 0.6 mg/kg of Dexamethasone Sodium Phosphate Injection 10mg/1ml given with equivalent volume of cherry syrup given orally once
  Dexamethasone Sodium Phosphate Injection
- Two Dose Dexamethasone: 0.6 mg/kg of Dexamethasone Sodium Phosphate Injection 10mg/1ml given with equivalent volume of cherry syrup given orally once in the Emergency Department (ED), followed by another dose of dexamethasone at home, which will be prescribed from the ED. The second dose will be the same dosage, but will be prescribed and may be pill or liquid form.
  Dexamethasone Sodium Phosphate Injection
Period: Overall Study
Arm/Group | Single Dose Dexamethasone | Two Dose Dexamethasone
Started | 154 | 154
Completed | 116 | 116
Not Completed | 38 | 38
Not completed — Lost to Follow-up | 25 | 27
Not completed — Given additional steroids with admission | 13 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Single Dose Dexamethasone | Two Dose Dexamethasone | Total
Number analyzed (Participants) | 116 | 116 | 232
Age, Continuous [Mean (Standard Deviation); unit: years] | 6.8 (3.9) | 8.2 (4.4) | 7.5 (4.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 44 | 92
  Male | 68 | 72 | 140
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 3
  Asian | 5 | 5 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 61 | 52 | 113
  White | 28 | 33 | 61
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 21 | 24 | 45
Tobacco exposure in home [Count of Participants; unit: Participants] | 32 | 31 | 63
Number of days with symptoms [Mean (Standard Deviation); unit: days] | 3.6 (9.7) | 3.1 (7.5) | 3.3 (8.7)
Current use of asthma controller medication [Count of Participants; unit: Participants] | 50 | 54 | 104
Number of previous hospital admissions [Mean (Standard Deviation); unit: admissions] | 1.4 (1.9) | 1.2 (2.5) | 1.3 (2.2)
Pediatric Asthma Score before albuterol administered [Mean (Standard Deviation); unit: PAS score] — Pediatric asthma Scores (based on respiratory rate by age, oxygen requirements, auscultation, retractions, dyspnea):
  5-7 Mild exacerbation 8-11 Moderate exacerbation 12-15 Severe exacerbation Population: PAS scores not available for all participants
  PAS score
    number analyzed (Participants) | 106 | 107 | 213
    (all) | 7.2 (1.8) | 6.9 (1.5) | 7.1 (1.6)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Returning to Care Following Discharge From the Emergency Department
Description: The investigators will determine if each patient had any unscheduled visits to the emergency room, urgent care or primary care physician.
Time Frame: 5 days
Measure: Count of Participants; unit: Participants
Arm/Group | Single Dose Dexamethasone | Two Dose Dexamethasone
Number analyzed (Participants) | 116 | 116
Participants | 14 | 12

2. Secondary Outcome: Reported Number of Days Until Symptom Resolution
Description: Will determine number of days to symptom resolution, including missed school days.
Time Frame: 5 days
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Single Dose Dexamethasone | Two Dose Dexamethasone
Number analyzed (Participants) | 116 | 116
Days | 2.4 (3.5) | 2.5 (3.4)

3. Other Pre Specified Outcome: Reported Side Effects Experienced by Participants
Description: The investigators will determine during phone follow up if patient experienced any side effects related to the Dexamethasone, including vomiting, mood swings, behavior changes, appetite changes, sweating or headache.
Time Frame: 5 days
Measure: Count of Participants; unit: Participants
Arm/Group | Single Dose Dexamethasone | Two Dose Dexamethasone
Number analyzed (Participants) | 116 | 116
Participants
  No side effects | 71 | 83
  Decreased Appetite | 4 | 7
  Difficulty Sleeping | 9 | 0
  Mood swings/Agitation | 7 | 3
  Headache | 3 | 1
  Other | 5 | 4
  Multiple | 17 | 18

ADVERSE EVENTS:
Time Frame: 5 days
Groups:
- Single Dose Dexamethasone: This group was the standard arm and received one single dose of dexamethasone in the Emergency department
- Two Doses of Dexamethasone: This group was the intervention group and received a dose of dexma
Arm/Group | Single Dose Dexamethasone | Two Doses of Dexamethasone
All-Cause Mortality (participants affected / at risk) | 0/116 | 0/116
Serious Adverse Events (participants affected / at risk) | 0/116 | 0/116
Other Adverse Events (participants affected / at risk) | 20/116 | 10/116
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Single Dose Dexamethasone (N=116) | Two Doses of Dexamethasone (N=116)
Decreased Appetite (Gastrointestinal disorders) | 4 | 7 — Reported decrease in appetite
Difficulty sleeping (General disorders) | 9 | 0 — Reported difficulty sleeping
Moodswing/Agitation (Psychiatric disorders) | 7 | 3 — Reported mood swings/agitation

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-11-09): https://cdn.clinicaltrials.gov/large-docs/27/NCT02192827/Prot_SAP_000.pdf
  • Informed Consent Form (2017-11-09): https://cdn.clinicaltrials.gov/large-docs/27/NCT02192827/ICF_001.pdf